CLINICAL TRIAL: NCT03434860
Title: Effect of Alive Multistrain Probiotic on Insulin Resistance in Type 2 Diabetes Patients
Brief Title: Effect of Probiotic on Insulin Resistance in Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Nazarii Kobyliak, Associate Professor of Endocrinology Department, PhD, Bogomolets National Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDO-4
Record Dates: First submitted 2018-01-21; First posted 2018-02-15 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Type2 Diabetes; Insulin Resistance; Probiotic
MeSH Terms: conditions — Insulin Resistance | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization was done by the study statistician based on a computer-generated list. The groups were homogeneous according to age, sex and diagnostic criteria. The assignment of groups was blind to participants, research staff and outcome assessors moreover, to maintain blind parallel study the statistician was not aware of the allocation of participants to intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- probiotic (Active Comparator): Over 8 weeks of interventional period, the patient received 1 sachet (10 grams) per day.
  Interventions: Dietary Supplement: probiotic
- placebo (Placebo Comparator): Over 8 weeks of interventional period, the patient received 1 sachet (10 grams) per day.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: probiotic — The multiprobiotic "Symbiter" which contains of 14 alive probiotic strains of Lactobacillus + Lactococcus (6×1010 CFU/g), Bifidobacterium (1×1010/g), Propionibacterium (3×1010/g), Acetobacter (1×106/g) genera. Over 8 weeks of interventional period, the patient received 1 sachet (10 grams) of probiotic per day.
  Arms: probiotic
Dietary Supplement: placebo — Over 8 weeks of interventional period, the patient received 1 sachet (10 grams) of gel per day
  Arms: placebo

SUMMARY:
Probiotics have beneficial effect on obesity related disorders in animal models. Despite a large number of animal data, randomized placebo-controlled trials (RCT) concluded that probiotics have a moderate effect on glycemic control-related parameters. However, effect of probiotics on insulin resistance are inconsistent. In this double-blind single center RCT, effect of alive multistrain probiotic vs. placebo on insulin resistance in type 2 diabetes patient will be assessed.

DETAILED DESCRIPTION:
In this single-center double blind, placebo controlled, parallel group study, type 2 diabetes patients from the Kyiv City Clinical Endocrinology Center will be selected. They will be randomly assigned to receive multiprobiotic "Symbiter" or placebo for 8-weeks administered as a sachet formulation in double-blind treatment. Randomization will be done by the study statistician based on a computer-generated list. The groups will be homogeneous according to age, sex and diagnostic criteria. The assignment of groups will be blind to participants, research staff and outcome assessors moreover, to maintain blind parallel study the statistician was not aware of the allocation of participants to intervention.

The multiprobiotic "Symbiter" will be supplied by Scientific and Production Company "O.D. Prolisok". It contains of 14 alive probiotic strains of Lactobacillus + Lactococcus (6×1010 CFU/g), Bifidobacterium (1×1010/g), Propionibacterium (3×1010/g), Acetobacter (1×106/g) genera. Over 8 weeks of interventional period, the patient received 1 sachet (10 grams) of probiotic and placebo per day. All sachets were identical with similar organoleptic characteristics (e.g., taste and appearance).

The pre-randomization period designed to minimize the effects of dietary changes on metabolic markers. For this purpose, 2 weeks before the study start, after inform consent signed, patients will be instructed in one-on-one sessions with a dietitian to follow a therapeutic lifestyle-change diet as classiﬁed by the NCEP. In addition, participants will be instructed to continue with stable anti-hyperglycemic treatment and received standardized mild physical training for 1 hour per day.

Patients who underwent study will be instructed to take the trial medication as prescribed. Throughout the study, weekly phone follow-up visits will be provided for assessment of compliance, adherence to the protocol, as well as the recording of adverse events. The effectiveness of therapy will be compared and evaluated separately in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* adult participants (ages 18-75, BMI ≥25 kg/m2) diagnosed with T2D according WHO (1999) for at least 6 months prior to the study;
* patient who treated with diet and exercise alone or metformin, SUs and insulin on a stabilized dose for at least 3 months before the study;
* presence of insulin resistance established as HOMA-IR≥2.0;
* HbA1c between 6.5 and 11.0 %;
* written informed consent.

Exclusion Criteria:

* presence of type 1 diabetes;
* treatment with other than mention in inclusion criteria antidiabetic drugs (pioglitazone, GLP-1 analogues, DPP IV inhibitors etc);
* regular use of a probiotic or prebiotic supplement within 3 months prior to enrollment;
* antibiotic use within 3 months prior to enrollment;
* uncontrolled cardiovascular or respiratory disease, decompensated liver disease including ascites, encephalopathy or variceal bleeding, active malignancy, or chronic infections;
* participation in other clinical trials;
* presence of pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2016-11-20 (Actual); Study Completion 2017-01-25 (Actual)

PRIMARY OUTCOMES:
HOMA-IR | 8 weeks compared to baseline
  HOMA-IR was calculated according to the formula: fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5

SECONDARY OUTCOMES:
HbA1c | 8 weeks compared to baseline
  HbA1c in %
fasting plasma insulins (FPI) | 8 weeks compared to baseline
  FPI in microU/L
fasting plasma glucose (FPG) | 8 weeks compared to baseline
  FPG in mmol/L
weight | 8 weeks compared to baseline
  weight in kg
waist circumferences (WC) | 8 weeks compared to baseline
  WC in cm
body mass index (BMI) | 8 weeks compared to baseline
  weight and height will be combined to report BMI in kg/m^2
cytokines levels | 8 weeks compared to baseline
  TNF-α, IL-1β, IL-6, IL-8, INF-γ

CONTACTS AND LOCATIONS:
Overall Officials: Petro Bodnar, Prof, Principal Investigator — Bogomolets National Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kobyliak N, Falalyeyeva T, Mykhalchyshyn G, Kyriienko D, Komissarenko I. Effect of alive probiotic on insulin resistance in type 2 diabetes patients: Randomized clinical trial. Diabetes Metab Syndr. 2018 Sep;12(5):617-624. doi: 10.1016/j.dsx.2018.04.015. Epub 2018 Apr 10. PMID 29661605